CLINICAL TRIAL: NCT03509064
Title: The Medico-economic Impact and Quality of Life of the Small-fiber Neuropathy Associated by Using Validated Scales (SF36, DN4, PROFAD SSI, ESPRI)
Brief Title: Medico-economic and Quality of Life Impact of Sjogren-associated Small Fiber Neuropathy
Acronym: SFINESS-QoLEco
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: LFB BIOMEDICAMENTS (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI17025J; 2017-A02858-45 (Other: IDRCB)
Record Dates: First submitted 2018-02-26; First posted 2018-04-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Primary Sjögren Syndrome; Small Fiber Neuropathy; Quality of Life; Medico-economic Impact
Keywords: Primary sjogren syndrome; Small fiber neuropathy; Quality of life; Medico-economic impact
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with small fiber neuropathy: patients with Sjogren syndrome have a definite small fiber neuropathy
  Interventions: Other: Collection sheet
- 2: Patients without peripheral neuropathy: patients with Sjogren syndrome without signs of peripheral neuropathy (small or large fiber)

INTERVENTIONS:
Other: Collection sheet — Using EQ5D questionnaire and a collection of care resources consumed by the patients during a period of 6 months associated by using validated scales (SF36, DN4, PROFAD SSI, ESPRI) : collection sheet
  Groups: 1: Patients with small fiber neuropathy

SUMMARY:
BACKGROUND Sjögren's syndrome is an autoimmune disease whose prevalence is estimated between 200 and 500 patients per 100,000 persons in France (120 to 500,000 patients). It affects women (90%) between 40 and 60 years of age and main manifestations are generalized sicca syndrome (ocular, oral, cutaneous) and arthralgia. In 20% of cases, Sjögren's syndrome is associated with peripheral neuropathies, and the most common form is painful small fiber neuropathy (SFN). SFNs are mainly featured by neuropathic pain including burns (90%), numbness (87.5%), tingling (72.5%), electric shocks (70%) and tingling (82.5%) and also autonomic disorders (50 to 70%).

However, there are still important issues that deserve to be investigated by clinical and basic research. Among these issues, this study will focus on:

* The impact of SFN on the quality of life of patients with Sjögren's syndrome.
* The medico-economic impact of the SFN taking into account the repercussions on the quality of life, including professional life, usual care cost (analgesics, medical and paramedical consultations, hospitalizations or emergency).

EXPECTED RESULTS

* Confirmation of the major impairment in the quality of life of patients with Sjogren-associated SFN
* Analysis of correlations to highlight or not clinical or biological factors associated with quality of life impairment.
* Evaluation of the cost attributed to the presence of an SFN in patients with Sjögren's syndrome and the pharmaco-economic interest of conventional therapeutic management (analgesic treatment, consultation pain) compared to the cost of more aggressive immunomodulatory treatments.

DETAILED DESCRIPTION:
Primary objective: Identify the predictors of quality of life impairment and costs of management of patients with Sjögren's syndrome and small fiber neuropathy (SFN).

Secondary objectives :

1. Hospital, drug and city-care costs
2. Distribution of cost items
3. Part of costs attributable to pSS-associated SFN
4. Loss of quality of life attributable to pSS-associated SFN
5. Relationship between the domains of the EQ 5D questionnaire and the other specific quality of life questionnaires
6. Association of the EQ 5D and other questionnaires with the costs (part of the costs variance that might be explained by the quality of life).

PATIENTS AND METHODS / Study population

Monocentric study in the Department of Internal Medicine of Lariboisière Fernand Widal Hospital.

All included patients fulfilled 2002-criteria of primary Sjogren syndrome.

Patients are classified into 2 arms:

Arm1: patients with Sjögren's syndrome and definite SFN

Arm2 ( Control Group) : patients with Sjögren's syndrome and WITHOUT clinical and paraclinical arguments for peripheral neuropathy

RESARCH PROCESS

This study will be based on the delivery and analysis of validated questionnaires (collection sheet) in chronic diseases, pains or Sjögren's syndrome:

* SF-36 for quality of life,
* DN4 questionnaire to estimate the probability of neuropathic pain
* EQ5D Health questionnaire
* ESSPRI (4 questions): Sjogren-patient questionnaire
* PROFAD-SSI (19 questions), to assess tiredness, discomfort, pain and dryness symptoms associated with Sjögren's syndrome.
* The economic evaluation will be done after the inclusion visit and will be based on the collection of care resources consumed by the patients during a period of 6 months

ELIGIBILITY:
Inclusion Criteria:

* Definite primary Sjögren syndrome
* Age over 18 years
* No biologics nor immunoglobulin therapy during the 6 months before study onset

Arm 1: patients with a small fiber neuropathy defined by the presence of a clinical AND one paraclinical abnormality

* (i) Clinical signs of small fibers involvement: thermo-algic sensory deficit or autonomic dysfunction or neuropathic pain with DN4 ≥4;
* AND
* (ii) Small fibers neurophysiological abnormalities (QST, laser evoked potentials, autonomic nervous system tests (sympathetic skin response test or Sudoscan®)
* OR
* (iii) abnormal intraepidermal nerve fiber density (skin biopsy)

Arm2 (control group): patients without signs of peripheral neuropathy (small or large fiber)

Exclusion Criteria:

* Presence of other causes of peripheral neuropathy

  * Acquired: Diabetes, AL amyloidosis, Alcoholism, celiac disease, Drugs, toxic, HIV, Sarcoidosis, systemic vasculitis, Guillain-Barré syndrome.
  * Hereditary: Transthyretin hereditary amyloidosis (TTR), hereditary sensory and autonomic neuropathy (HSAN), Fabry's disease
* Patients with impaired thermo-algic sensitivity and / or dysautonomia and / or pain with DN4 ≥ 4 AND normal diagnostic tests (normal neurophysiological tests AND normal skin biopsy) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included patients fulfilled 2002-criteria of primary Sjogren syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Measure of quality of life impairment by SF 36 scale | Month 3
  For each of the eight domains that the SF36 measures an aggregate percentage score is produced. The percentage scores range from 0% (lowest or worst possible level of functioning) to 100% (highest or best possible level of functioning).
  It easy to set up a computerised database (e.g., in MS Excel or similar) to calculate the percentages and averages

SECONDARY OUTCOMES:
Hospitalization costs' | during a period of 6 months
  using a collection sheet
Drug costs' | during a period of 6 months
  using a collection sheet
City care costs' | during a period of 6 months
  using a collection sheet
Distribution of cost items | during a period of 6 months
  using a collection sheet
Part of costs attributable to primary Sjögren syndrome-associated small fiber neuropathy. | during a period of 6 months
  using a collection sheet
Loss of quality of life attributable to primary Sjögren syndrome-associated small fiber neuropathy. | during a period of 6 months
  The loss of quality of life is appreciated by using a collection sheet (detailed in the research process)
Evaluation of the domains of the EQ 5D questionnaire | during a period of 6 months
  using a collection sheet
Evaluation of specific quality of life questionnaire | during a period of 6 months
  using a collection sheet

CONTACTS AND LOCATIONS:
Overall Officials: Damien SÈNE, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département de Médecine Interne - Hôpital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided